CLINICAL TRIAL: NCT05899231
Title: OPAL: Online Prehabilitation for Patients Awaiting Liver Transplantation - a Multicenter Randomized Controlled Trial to Reduce Physical Frailty and Improve Health Outcomes
Brief Title: Online Prehabilitation for Patients Awaiting Liver Transplantation
Acronym: OPAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00125367
Record Dates: First submitted 2023-05-15; First posted 2023-06-12 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Cirrhosis, Liver; Liver Transplant Surgery; Liver Disease
Keywords: frailty; transplant; nutrition; exercise; ehealth; application; wellness; prehabilitation; sarcopenia; malnutrition; physical function; digital; virtual; online
MeSH Terms: conditions — Liver Cirrhosis; Liver Diseases; Frailty; Motor Activity; Sarcopenia; Malnutrition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation Group (Experimental): The prehabilitation group will be provided with access to the online digital web platform which contains the weekly acceptance and commitment therapy based education videos, nutrition intervention, and exercise intervention.
  Interventions: Behavioral: Prehabilitation Programming
- Usual Care (No Intervention): This group will receive standard care for LT candidates with cirrhosis and will be provided with standard online exercise, nutrition, and behavioural resources. Control participants will not receive access to the online digital platform.

INTERVENTIONS:
Behavioral: Prehabilitation Programming — 12-weeks of online prehabilitation programming including:
  1.12 weeks of nutrition programming focused on achieving a guideline- based protein intake of 1.2-1.5 g/kg/day. Participants will participate in a dietitian assessment and 0-2 dietitian follow-ups stratified by risk and 5 virtual group nutrition classes. Participants will be provided with a whey protein powder supplement - dosing stratified by risk.
  2.10 weeks of exercise programming focused on completion of 3 full- body resistance/aerobic exercise sessions weekly (1 or 2 virtual group classes as per patient preference + 1 or 2 pre-recorded home exercise videos).
  3.12 weeks of acceptance and commitment therapy based educational videos and online activities focused on reducing stress and anxiety and improving motivation and adherence.
  Arms: Prehabilitation Group

SUMMARY:
Physical frailty is common in patients awaiting liver transplantation and has been associated with poor health outcomes. There is promising data from small studies showing that behavioural, nutrition, exercise therapy (prehabilitation) improves physical function in patients while they are waiting for a liver transplant.

The proposed trial will assess if a 12-week online prehabilitation program improves physical function in patients listed for liver transplantation. Over 4 years, 177 patients will be recruited from 6 transplant centres across Canada and will be randomized to receive either the online prehabilitation program or usual care.

The primary outcome of physical function will be evaluated using the FTSST at baseline and 12 weeks (or last timepoint before transplant) assessed virtually or in-person. Secondary outcomes include liver specific physical frailty, aerobic fitness, health-related quality of life (QoL), participant experience and acceptability. Exploratory outcomes include other virtual and in-person physical function measures, covert hepatic encephalopathy (CHE), sarcopenia, malnutrition, adherence, behaviour factors, clinical and post-transplant outcomes. Results will be compared between the intervention and usual care groups.

DETAILED DESCRIPTION:
This multi-centre randomized controlled trial (RCT) will be completed across the six major LT programs in Canada: Vancouver, Edmonton, Calgary, Toronto, London, and Montreal.

Participants involved in this study will be LT transplant candidates with cirrhosis who are receiving care at one of the six participating LT programs.

Participants will be assessed for eligibility, provided informed signed consent, complete baseline testing and then be randomized to the prehabilitation arm or usual care. Participants will be randomized in a 2:1 ratio between groups.

Prehabilitation Arm:

The 12 week prehabilitation program includes exercise, nutrition and psychological components that is accessed through the online digital web platform.

* The nutrition program includes a nutritional assessment, provision of a daily protein intake target (1.2-1.5 g/kg/day), online group sessions, and follow ups. Participants will also be provided with a clinically tested whey protein powder supplement with dosage based on their malnutrition scoring done at baseline. Follow ups will also be provided based on malnutrition scoring done at baseline.
* The exercise program includes an exercise assessment, follow along exercise videos, and weekly virtual live exercise sessions. The exercise specialist will advise one of three levels of exercise programming for each participant. Participants will be advised to complete 3 exercise sessions weekly from a combination of virtual group sessions and follow along videos and to participate in planned aerobic activity as much as possible.
* The weekly acceptance and commitment therapy based educational videos focus on reducing stress and anxiety and improving motivation and adherence.

Control/Usual Care Arm:

This group will receive standard care for LT candidates with cirrhosis and will be provided with standard online exercise, nutrition, and behavioural resources. Control participants will not receive access to the online digital platform. A short questionnaire will be sent to control participants every 4 weeks to track changes in physical activity.

Post-Transplant follow-up In the subgroup of patients who undergo LT, the same in-person and virtual testing will be carried out at 12 weeks post-transplant (timing may vary due to site clinic flow)

Data Collection Plan

Sample size calculations are based on the primary outcome (the chair stand test: time to complete 5 sit-to-stands) using individual data from our local exercise study in cirrhosis (n=59), plus our sit-to-stand data from our study of 694 patients. After accounting for lack of trial completion, loss to follow up, the total sample size is 177, with 59 participants in the control and 118 in the intervention arm.

1. Quantitative outcomes: Baseline and primary/secondary/exploratory outcome data will be collected with in-person and/or virtual visits at baseline, week 12 (end of trial) and 12 weeks post-transplant (in the subgroup of patients who undergo LT). Charts will be reviewed for information on death, hospitalization, ambulatory care visits, medications and transplantation for up to 2 years after randomization in all participants. Dietary intake data (24-hour recall) may be collected using third party software.
2. Qualitative data: Interviews/Focus groups will be conducted at the end of the study in a virtual format. Participation in the interviews/focus groups will be optional.

Types of analyses

1. Quantitative outcomes: Baseline demographic and clinical characteristics will be compared between groups to identify differences that may exist despite randomization. Continuous variables will be screened for assumptions of normality, and descriptive analyses will be presented for participant demographics, medical and outcome variables. Sex will be used in subgroup analysis of primary and secondary outcomes. It will also be a covariate for exploratory analysis in corresponding models. All analyses will adhere to the intention-to-treat principle.
2. Qualitative data: Qualitative data will be analyzed inductively following a theoretical thematic approach. Data will be coded, with codes combined into larger categories and theme, with the goal of highlighting participant experiences and acceptability (barriers, facilitators) of the OPAL platform and intervention. Data collection and analysis will occur concurrently in order to enable refinement of interview/focus guide questions and deeper exploration of emerging themes.

Primary outcome: The primary outcome (sit to stand test; time to do 5 sit-to-stands) will be analyzed by linear mixed models with random effects, adjusted for baseline score as a covariate. Sites will be entered as random effects.

Secondary/exploratory outcomes: (1) Quantitative outcomes: Similar types of models will be used for continuous secondary/exploratory outcomes. To examine predictors of exercise and nutrition adherence (e.g. COM-B results), generalized linear models with binary outcome will be employed. To evaluate the potential effect of selected demographic variables on outcomes, as an exploratory analysis, models will be adjusted for clinically significant variables (e.g. sex, gender, digital technology proficiency). Results will be primarily descriptive. Exploratory per-protocol analysis will be performed, and the results will be presented if substantial differences are found between this group and the intention-to-treat group.

ELIGIBILITY:
Inclusion Criteria:

≥18 years old with cirrhosis (confirmed with transient elastography by FibroScan, histology, or imaging-based assessment with compatible clinical picture), referred for transplant and are assessed to have a high likelihood of being listed according to a preliminary review by hepatologist or are already listed for LT, are pre-frail or frail on the liver frailty index (LFI) or (added August 30, 2024) pre-frail or frail on the TeLeFI (prefrail LFI 3.2-4.3 and frail LFI ≥4.4), have English or French language proficiency, and own an internet-connected device.

Exclusion Criteria:

* Listed for living related donor transplantation with expected time on the wait list <12 weeks, or model for end-stage liver disease (MELD-Na) Score >26 (Justification: time to transplant is very short)
* Robust status on frailty testing (LFI 0-3.1) (Justification: unlikely to see benefit)
* Unable to provide informed consent
* Presence of a clinical condition that makes the intervention unsafe or infeasible (e.g. unable to follow instruction) or unsafe environment for virtual participation
* Life expectancy less than 6 months, compassionate care (clinician judgment) (Justification: unlikely to see benefit)
* Recent variceal bleed or history of varices not on adequate prophylaxis (Justification: acute exercise increases portal pressure
* Transplant indication is cholangiocarcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in time to do 5-sit-to-stands from baseline | Week 0
  A time to complete 5 chair stands of >15 seconds predicts morbidity and mortality in patients with cirrhosis. This test shows promise as a frailty measure that could be evaluated over a virtual platform
Change in time to do 5-sit-to-stands from baseline | Week 12
  A time to complete 5 chair stands of >15 seconds predicts morbidity and mortality in patients with cirrhosis. This test shows promise as a frailty measure that could be evaluated over a virtual platform

SECONDARY OUTCOMES:
Change in liver frailty index from baseline | Week 0
  Liver frailty will be assessed with a cirrhosis-specific tool. The in-person LFI which includes grip strength, chair stand and balance testing, or the virtual TeLeFI which includes virtual FTSST, three stance balance test, and selected questions from validated surveys. The LFI is an independent predictor of waitlist mortality and hospitalization.
  The LFI score can be calculated using an online calculator (available at http://liverfrailtyindex.ucsf.edu), with patient physical frailty categorized as robust, prefrail, and frail according to their index (index < 3.2, robust; 3.2-4.5, prefrail; and >4.5, frail).
  Higher scores mean a worse outcome.
Change in liver frailty index from baseline | Week 12
  Liver frailty will be assessed with a cirrhosis-specific tool. The in-person LFI which includes grip strength, chair stand and balance testing, or the virtual TeLeFI which includes virtual FTSST, three stance balance test, and selected questions from validated surveys. The LFI is an independent predictor of waitlist mortality and hospitalization.
  The LFI score can be calculated using an online calculator (available at http://liverfrailtyindex.ucsf.edu), with patient physical frailty categorized as robust, prefrail, and frail according to their index (index < 3.2, robust; 3.2-4.5, prefrail; and >4.5, frail).
  Higher scores mean a worse outcome.
Changes in virtual physical function testing over time (2-min step test) | Week 0
  The 2-min step test is used to assess aerobic endurance and functional fitness. The subject marches in place for two minutes.
  The literature supports good correlation of this virtual measure when compared to in-person testing
Changes in virtual physical function testing over time (2-min step test) | Week 12
  The 2-min step test is used to assess aerobic endurance and functional fitness. The subject marches in place for two minutes.
  The literature supports good correlation of this virtual measure when compared to in-person testing
Change in health-related quality of life from baseline (CLDQ) | Week 0
  The disease-specific Chronic Liver Disease Questionnaire (CLDQ) is validated in cirrhosis.
  Overall CLDQ scores calculated for each domain range from 1 (most impaired) to 7, with higher scores indicating a minimum frequency of symptoms and hence a better HRQOL.
Change in health-related quality of life from baseline (CLDQ) | Week 12
  The disease-specific Chronic Liver Disease Questionnaire (CLDQ) is validated in cirrhosis.
  Overall CLDQ scores calculated for each domain range from 1 (most impaired) to 7, with higher scores indicating a minimum frequency of symptoms and hence a better HRQOL.
Change in health-related quality of life from baseline (EQ5D5L and EQVAS) | Week 0
  The EuroQoL 5-D-5L and visual analog scale (EQ-VAS) are generic tools also validated in LT candidates and recipients.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Change in health-related quality of life from baseline (EQ5D5L and EQVAS) | Week 12
  The EuroQoL 5-D-5L and visual analog scale (EQ-VAS) are generic tools also validated in LT candidates and recipients.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Qualitative Acceptability Data | Week 12
  Inductive analysis of post-trial semi-structured interviews/focus groups with participants

OTHER OUTCOMES:
Change in time to do 5-sit-to-stands from baseline | Week 8
  A time to complete 5 chair stands of >15 seconds predicts morbidity and mortality in patients with cirrhosis. This test shows promise as a frailty measure that could be evaluated over a virtual platform
  Completed at week 8 to account for the possibility of transplantation or loss-to-follow-up before the end of the 12 weeks.
Change in sarcopenia from baseline | Week 0
  Calf circumference is a simple measure for appendicular skeletal muscle and predicting sarcopenia
Change in sarcopenia from baseline | Week 12
  Calf circumference is a simple measure for appendicular skeletal muscle and predicting sarcopenia
Change in distance in the 6 minute walk test from baseline | Week 0
  6MWT distance correlates with waitlist mortality and QoL and is recommended by the American Society of Transplantation. It is associated with protein intake, activity level and physical function/ frailty.
Change in distance in the 6 minute walk test from baseline | Week 12
  6MWT distance correlates with waitlist mortality and QoL and is recommended by the American Society of Transplantation. It is associated with protein intake, activity level and physical function/ frailty.
Change in covert hepatic encephalopathy from baseline | Week 0
  The EncephalApp Stroop (Stroop) test is a reliable, easy-to-use diagnostic test for CHE. It evaluates psychomotor speed and cognitive flexibility.
Change in covert hepatic encephalopathy from baseline | Week 12
  The EncephalApp Stroop (Stroop) test is a reliable, easy-to-use diagnostic test for CHE. It evaluates psychomotor speed and cognitive flexibility.
Change in health-related quality of life from baseline (EQ5D5L and EQVAS) | Week 8
  The EuroQoL 5-D-5L and visual analog scale (EQ-VAS) are generic tools also validated in LT candidates and recipients.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Change in health-related quality of life from baseline (CLDQ) | Week 8
  The disease-specific Chronic Liver Disease Questionnaire (CLDQ) is validated in cirrhosis.
  Overall CLDQ scores calculated for each domain range from 1 (most impaired) to 7, with higher scores indicating a minimum frequency of symptoms and hence a better HRQOL.
Change in 6-item COM-B scale over time during intervention | Week 4
  Perceived capability, opportunity, and motivation will be assessed over the trial period to understand how the COM-B impacts adherence. Each item is scaled (0 [strongly disagree] to 7 [strongly agree]) and 3 subscores are computed. A higher score means higher perceived capability, opportunity, and motivation
Change in 6-item COM-B scale over time during intervention | Week 8
  Perceived capability, opportunity, and motivation will be assessed over the trial period to understand how the COM-B impacts adherence. Each item is scaled (0 [strongly disagree] to 7 [strongly agree]) and 3 subscores are computed. A higher score means higher perceived capability, opportunity, and motivation
Change in 6-item COM-B scale over time during intervention | Week 12
  Perceived capability, opportunity, and motivation will be assessed over the trial period to understand how the COM-B impacts adherence. Each item is scaled (0 [strongly disagree] to 7 [strongly agree]) and 3 subscores are computed. A higher score means higher perceived capability, opportunity, and motivation.
Change in health-related quality of life from baseline (EQ5D5L and EQVAS) | Post-transplant (12 weeks after transplant date)
  The EuroQoL 5-D-5L and visual analog scale (EQ-VAS) are generic tools also validated in LT candidates and recipients.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Change in health-related quality of life from baseline (CLDQ) | Post-transplant (12 weeks after transplant date)
  The disease-specific Chronic Liver Disease Questionnaire (CLDQ) is validated in cirrhosis.
  Overall CLDQ scores calculated for each domain range from 1 (most impaired) to 7, with higher scores indicating a minimum frequency of symptoms and hence a better HRQOL.
Changes in virtual physical function testing over time (Single leg balance test) | Week 0
  The single leg balance test is used to assess static postural and balance control. The test assesses the length of time the subject can maintain their balance
  The literature supports good correlation of this virtual measure when compared to in-person testing
Changes in virtual physical function testing over time (Single leg balance test) | Week 8
  The single leg balance test is used to assess static postural and balance control. The test assesses the length of time the subject can maintain their balance
  The literature supports good correlation of this virtual measure when compared to in-person testing
Changes in virtual physical function testing over time (Single leg balance test) | Week 12
  The single leg balance test is used to assess static postural and balance control. The test assesses the length of time the subject can maintain their balance
  The literature supports good correlation of this virtual measure when compared to in-person testing
Changes in virtual physical function testing over time (Single leg balance test) | Post-transplant (12 weeks after transplant date)
  The single leg balance test is used to assess static postural and balance control. The test assesses the length of time the subject can maintain their balance
  The literature supports good correlation of this virtual measure when compared to in-person testing
Changes in virtual physical function testing over time (2-min step test) | Week 8
  The 2-min step test is used to assess aerobic endurance and functional fitness. The subject marches in place for two minutes.
  The literature supports good correlation of this virtual measure when compared to in-person testing
Changes in virtual physical function testing over time (2-min step test) | Post-transplant (12 weeks after transplant date)
  The 2-min step test is used to assess aerobic endurance and functional fitness. The subject marches in place for two minutes.
  The literature supports good correlation of this virtual measure when compared to in-person testing
Number of participants who died during the 12 week trial | Week 12
  Death will be collected through chart review
Number of hospitalizations and ambulatory clinic visits during the 12 week trial | Week 12
  Hospitalizations and ambulatory clinic visits will be collected through chart review
Number of participants who were transplanted during the 12 week trial | Week 12
  Data on transplantations occurring during the trial will be collected through chart review
Number of participants who died during the 2 years post-study completion | 2 years post-study completion
  Death will be collected through chart review. Consent will be obtained to extend this to 2 years of extended follow-up for all participants and to link to administrative data-repositories for follow-on research.
Number of hospitalizations and ambulatory clinic visits during the 2 years post-study completion | 2 years post-study completion
  Hospitalizations and ambulatory clinic visits will be collected through chart review. Consent will be obtained to extend this to 2 years of extended follow-up for all participants and to link to administrative data-repositories for follow-on research.
Number of participants who were transplanted during the 2 years post-study completion | 2 years post-study completion
  Data on transplantations occurring during the trial will be collected through chart review. Consent will be obtained to extend this to 2 years of extended follow-up for all participants and to link to administrative data-repositories for follow-on research.
Economic Evaluation | Week 12
  Healthcare access and hospital usage will be collected through patient survey.
Total Length of stay at time of transplant | Post-transplant up to 3 months of the trial data collection period
  In participants transplanted within 3 months of the end of the trial data collection period, we will ascertain total length of stay at time of transplant
Intensive care unit length of stay at time of post transplant | Post-transplant up to 3 months of the trial data collection period
  In participants transplanted within 3 months of the end of the trial data collection period, we will ascertain intensive care unit length of stay
Days of mechanical ventilation at time of post transplant | Post-transplant up to 3 months of the trial data collection period
  In participants transplanted within 3 months of the end of the trial data collection period, we will ascertain days of mechanical ventilation
Discharge location from hospital at time of transplant | Post-transplant up to 3 months of the trial data collection period
  In participants transplanted within 3 months of the end of the trial data collection period, we will ascertain discharge home from hospital (versus rehabilitation, nursing home or other institutional location)
Readmissions within 30 days at time of transplant | Post-transplant up to 3 months of the trial data collection period
  In participants transplanted within 3 months of the end of the trial data collection period, we will ascertain any readmissions within 30 days.
Malnutrition | Week 0
  The Patient-Generated Subjective Global Assessment (PG-SGA) is an instrument for assessment of nutrition status in patients with cancer and other diseases. It contains both a patient and a practitioner section. A higher score means worse outcomes.
  The numerical PG-SGA score provides professionals with clearer guidelines as to the level of medical nutrition therapy needed in a given case, while the A, B, or C rating provides an overall picture of a patient's current status. (A = well nourished, B = moderately malnourished or suspected malnutrition and C = severely malnourished).
Malnutrition | Week 12
  The Patient-Generated Subjective Global Assessment (PG-SGA) is an instrument for assessment of nutrition status in patients with cancer and other diseases. It contains both a patient and a practitioner section. A higher score means worse outcomes.
  The numerical PG-SGA score provides professionals with clearer guidelines as to the level of medical nutrition therapy needed in a given case, while the A, B, or C rating provides an overall picture of a patient's current status. (A = well nourished, B = moderately malnourished or suspected malnutrition and C = severely malnourished).
Adverse events | Week 12
  Major: death or hospitalization for an event occurring during or up to 3 h after exercise; cardiovascular events (stroke, myocardial infarction); permanent disability; angina, syncope, arrhythmia; variceal bleeding. Minor: hypoglycemia, hyper- or hypotension requiring medical attention, musculoskeletal injury or fall.
Changes in health care provider support from baseline | Week 0
  Chart review will record days of enteral or parenteral nutrition provided during hospitalization or as an outpatient and will also record exposure to the number of non-intervention digital platform based exercise sessions attended through to end of extended follow-up.
Changes in physical activity levels from baseline | Week 0
  Participants will be asked to journal about the amount of exercise they take part in over the course of the 12 week trial and for as long as possible into the extended follow-up period as they are willing to.
Changes in health care provider support from baseline | Week 4
  Chart review will record days of enteral or parenteral nutrition provided during hospitalization or as an outpatient and will also record exposure to the number of non-intervention digital platform based exercise sessions attended through to end of extended follow-up.
Changes in physical activity levels from baseline | Week 4
  Participants will be asked to journal about the amount of exercise they take part in over the course of the 12 week trial and for as long as possible into the extended follow-up period as they are willing to.
Changes in health care provider support from baseline | Week 8
  Chart review will record days of enteral or parenteral nutrition provided during hospitalization or as an outpatient and will also record exposure to the number of non-intervention digital platform based exercise sessions attended through to end of extended follow-up.
Changes in physical activity levels from baseline | Week 8
  Participants will be asked to journal about the amount of exercise they take part in over the course of the 12 week trial and for as long as possible into the extended follow-up period as they are willing to.
Changes in health care provider support from baseline | Week 12
  Chart review will record days of enteral or parenteral nutrition provided during hospitalization or as an outpatient and will also record exposure to the number of non-intervention digital platform based exercise sessions attended through to end of extended follow-up.
Changes in physical activity levels from baseline | Week 12
  Participants will be asked to journal about the amount of exercise they take part in over the course of the 12 week trial and for as long as possible into the extended follow-up period as they are willing to.
Changes in functional status from baseline | Week 0
  The TeLeFI assesses frailty and functional status virtually via phone and/or video capability without specialized equipment to identify patients who may be at risk of frailty as defined by the in-person LFI
Changes in functional status from baseline | Week 8
  The TeLeFI assesses frailty and functional status virtually via phone and/or video capability without specialized equipment to identify patients who may be at risk of frailty as defined by the in-person LFI
Changes in functional status from baseline | Week 12
  The TeLeFI assesses frailty and functional status virtually via phone and/or video capability without specialized equipment to identify patients who may be at risk of frailty as defined by the in-person LFI
Adherence to prehabilitation program goals | Week 12
  (i) 70% adherence to target protein intake and protein powder supplementation (assessed by dietary intake, nutrition check ins, platform metrics and monthly nutrition questionnaires), (ii) 70% adherence to exercise sessions (assessed by attendance, check ins, platform metrics) excluding study weeks with interruptions to programming due to health related issues (e.g. transplant dry runs, hospital admissions as these are common in patients awaiting LT)

CONTACTS AND LOCATIONS:
Overall Officials: Puneeta Tandon, Principal Investigator — University of Alberta
Locations (6):
- Canada (6):
  - Foothills Medical Centre, Calgary, Alberta
  - Kaye Edmonton Clinic, Edmonton, Alberta
  - Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Toronto General Hospital - Ajmera Transplant Centre, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No